CLINICAL TRIAL: NCT02891655
Title: KERatoconus and Metalloproteinases InvesTigation
Acronym: KERMIT
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: EGN_2016_6
Record Dates: First submitted 2016-08-25; First posted 2016-09-07 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- surgery for keratoconus
  Interventions: Other: immuno-histo-chemical analysis
- refractive surgery (control patients)
  Interventions: Other: immuno-histo-chemical analysis

INTERVENTIONS:
Other: immuno-histo-chemical analysis — in vitro immuno-histo-chemical analysis of corneal epithelium

SUMMARY:
Corneal stromal thinning observed in keratoconic eyes could result from an increased synthesis of MMP at the level of the anterior stroma and the corneal epithelium induced by an overexpression of the Extracellular Matrix Metalloproteinase Inducer (EMMPRIN) and Galectin-3 by epithelial cells. A differential expression of EMMPRIN, Galectin-3 and metalloproteinases (MMP) may be observed between the apex of the keratoconus and the peripheral cornea. Highlighting the implication of EMMPRIN and Galectin-3 could lead to the development of specific inhibitors to slow or to stop keratoconus evolution.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* Patient with keratoconus undergoing corneal collagen cross-linking (epithelium-off methods)
* Patient with keratoconus undergoing his first corneal graft for optical indication (control)

Exclusion Criteria:

* Patient with keratoconus undergoing corneal graft for tectonic indication
* Patient undergoing corneal refractive surgery (refractive photokeratectomy) with a normal topography, a normal slit lamp examination and no previous ophthalmic condition (control)
* pregnant or breast feeding patient
* patient under judiciary protection
* patient opposition to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with keratoconus and controls subjects without keratoconus
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2016-12-02 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-11-26 (Actual)

PRIMARY OUTCOMES:
expression of the Extracellular Matrix Metalloproteinase Inducer (EMMPRIN) in epithelial cells | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Eric GABISON, MD, PhD, Principal Investigator — Fondation OPH A de Rothschild
Locations (1):
- Fondation Opthalmologique A de Rothschild, Paris, France